CLINICAL TRIAL: NCT05543707
Title: A Phase 2 Double-blind, Randomized Study to Evaluate the Antiviral Activity, Safety, and Efficacy of Orally Administered PBI-0451(Pomotrelvir) Compared With Placebo in Nonhospitalized Symptomatic Adults With COVID-19
Brief Title: PBI-0451 (Pomotrelvir) Phase 2 Study in Nonhospitalized Symptomatic Adults With COVID-19
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim analysis concluded primary endpoint was not met
Sponsor: Pardes Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PBI-0451-0002; 2022-001195-33 (EudraCT Number)
Record Dates: First submitted 2022-09-07; First posted 2022-09-16 (Actual); Results first posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-08

CONDITIONS: COVID-19
Keywords: COVID; SARS-CoV-2; Coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — PBI-0451; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PBI-0451 (Pomotrelvir) (Experimental): PBI-0451(Pomotrelvir): 2 x 350 mg tablets administered orally twice daily (BID) (1400 mg/day) with food for 5 days (10 total doses)
  Interventions: Drug: PBI-0451 (Pomotrelvir)
- Placebo (Placebo Comparator): PBI-0451(Pomotrelvir): 2 x placebo to match PBI-0451(Pomotrelvir) tablets administered orally twice daily (BID) with food for 5 days (10 total doses)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PBI-0451 (Pomotrelvir) — 2 × 350 mg tablets administered orally twice daily (BID) (1400 mg/day) with food for 5 days (10 total doses)
  Other Names: Active
  Arms: PBI-0451 (Pomotrelvir)
Drug: Placebo — 2 × placebo to match PBI-0451(Pomotrelvir) tablets administered orally BID with food for 5 days (10 total doses)
  Arms: Placebo

SUMMARY:
This is a phase 2 double-blind, randomized study of PBI-0451(Pomotrelvir) in nonhospitalized symptomatic adults with COVID-19. PBI-0451(Pomotrelvir) is a new chemical entity and inhibitor of the main protease of coronaviruses, including the SARS-CoV-2 that causes COVID-19 disease. This study is designed to evaluate the antiviral activity, safety, and efficacy of orally administered PBI-0451(Pomotrelvir) compared with placebo.

DETAILED DESCRIPTION:
Following randomization on Day 1, subjects will complete baseline assessments prior to receiving their first dose of study drug (PBI-0451 or placebo).

Randomization will be stratified as follows:

* SARS-CoV-2 positive direct test diagnosis ≤ 3 days (target 30%) versus > 3 days from first onset of COVID-19 symptom(s) ≤ 5 days prior to randomization
* Received primary vaccination series, alone versus any booster shots
* PK substudy participation versus nonparticipation Study drug will be taken with food, approximately 12 hours between doses, at approximately the same time for each BID dose for the remainder of the 5 days of treatment.All subjects will have additional safety and efficacy assessments during the 28-day study period. A follow-up visit (eg, telephone visit, virtual visit, clinic visit, etc. as convenient) will be conducted at Week 24 (± 20 days) after the last dose of study drug for all subjects. Information regarding ongoing or recurrent COVID-19 symptoms, survival status, pregnancy status (for female subjects of childbearing potential and female partners of male subjects), and any hospitalizations or acute/critical care visits (eg, non-admitted hospital or other care facility)that have occurred since the last study visit will be collected. A team of medically qualified individuals, including but not limited to, the Sponsor and the CRO Medical Monitors, and the Drug Safety Consultant are responsible for ongoing review of all AEs, concomitant medications, laboratory values (including virology), and vital signs (including pulse oximetry), worsening of symptoms (COVID-19 symptom questionnaire, including dyspnea), acute/critical care visits (eg, nonadmitted hospital or other care facility), and study drug discontinuations, at a minimum monthly basis throughout the study, per the Safety Monitoring Plan. Subjects who experience severe COVID-19 illness (defined in this study as sustained pulse oximetry <94%, a respiratory rate of >30 breaths/min, or dyspnea that requires medical attention) should discontinue study drug and be immediately referred by the Investigator to emergency care or treated by the Investigator for standard of care treatment of symptoms including, but not limited to, other antivirals, supplemental oxygen, corticosteroids, Janus kinase inhibitors, or interleukin-6 blockers, in accordance with the NIH Treatment Guidelines (NIH 2022). The subject should continue participation in the study, with study drug discontinued, for safety follow-up and clinical outcome of the medically attended visit.

ELIGIBILITY:
Inclusion Criteria:

1. Can understand and sign a written informed consent form (ICF), which must be obtained prior to initiation of any study procedures.
2. Onset of COVID-19 symptoms ≤ 5 days prior to randomization with a positive SARS-CoV-2 test ≤ 24 hours prior to randomization. Authorized NAAT or antigen tests that detect viral RNA or protein, respectively, are allowed.
3. Received primary vaccination series as defined by Centers for Disease Control and Prevention (CDC). Subjects should be advised during informed consent that alternate therapies may be available outside of study participation.
4. ≥ 2 symptoms of acute COVID-19 infection as determined by the investigator from the symptoms listed on the COVID-19 symptoms questionnaire present at randomization
5. Male and nonpregnant, nonlactating female subjects 18 to < 65 years of age. Females must have a negative serum or urine pregnancy test at screening and prior to the first dose of study drug unless permanently sterile or in a postmenopausal state (see Appendix 3).
6. Male and female subjects and/or their heterosexual partners must either be of nonchildbearing potential or must use effective contraception from screening through 90 days after the last dose of study drug (see Appendix 3)
7. Female subjects must refrain from egg donation and in vitro fertilization during treatment and for ≥ 28 days after the last dose of study drug
8. Male subjects must refrain from sperm donation from screening through 90 days after the last dose of study drug
9. Normal 12-lead electrocardiogram (ECG) evaluation without clinically significant abnormalities
10. Able and willing to comply with all study requirements

Exclusion Criteria:

1. Considered at high-risk of developing severe illness from COVID-19 defined as ≥ 1 CDC underlying medical condition associated with an increased risk of developing severe illness from COVID-19 (see Appendix 5)
2. Unvaccinated against SARS-CoV-2 (defined as having not completed a primary vaccination series)
3. Any SARS-CoV-2 vaccination within 3 month prior to randomization or anticipated to receive a SARS-CoV-2 vaccination (including a booster) during the 28-day study period
4. Currently hospitalized or expected to require hospitalization for COVID-19 within 48 hours of randomization
5. Currently being treated or expected to be treated for COVID-19 with monoclonal antibodies, convalescent serum, or direct-acting antiviral agents (all potential subjects should be informed of evolving treatment options during informed consent that alternate therapies may or may not be available to them outside of study participation)
6. Any clinical condition or laboratory result considered by the investigator to indicate any unstable or poorly controlled underlying clinically significant medical condition(s), active disseminated infection (other than SARS-CoV-2), or other medical condition that could represent a risk to the subject, including increasing the likelihood of a safety event, affect subject compliance, or affect efficacy and/or safety data collected during the 28-day study period
7. Known active liver disease, including nonalcoholic steatohepatitis/nonalcoholic fatty liver disease, chronic or active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection, primary biliary cirrhosis, Child-Pugh Class B or C, chronic alcoholic liver disease, or acute liver failure
8. Receiving dialysis or having known severe renal impairment (chronic kidney disease, Stage 4 or above)
9. Unable or unwilling to comply with the protocol procedures
10. Participating in another interventional study with an investigational compound or device, including those for COVID-19
11. Known prior participation in this study or another study involving PBI-0451(Pomotrelvir)
12. Females who are pregnant or breastfeeding
13. Oxygen saturation of < 94% on room air

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 242 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Wilfret, MD, Study Director — Pardes Biosciences
Locations (54):
- United States (54):
  - Voyage Medical, Mesa, Arizona
  - Franco A Felizarta MD, Bakersfield, California
  - Hope Clinical Research, LLC, Canoga Park, California
  - Biopharma Informatic, LLC, Encino, California
  - Ascada Research LLC, Fullerton, California
  - Ark Clinical Research - Long Beach - Clinedge - PPDS, Long Beach, California
  - Valiance Clinical Research, Tarzana, California
  - Allianz Research Institute - Colorado, Westminster, California
  - TrueBlue Clinical Research- Brandon - HyperCore - PPDS, Brandon, Florida
  - Beautiful Minds Clinical Research Center, Cutler Bay, Florida
  - Indago Research and Health Center, Hialeah, Florida
  - Quality Research of South Florida, Hialeah, Florida
  - Gonzalez M.D. & Aswad M.D. Health Care Services, Miami, Florida
  - Universal Medical and Research Center, LLC, Miami, Florida
  - CCM Clinical Research Group, Miami, Florida
  - D&H National Research Centers, Miami, Florida
  - Allied Biomedical Research Institute, Miami, Florida
  - Florida International Medical Research, Miami, Florida
  - P&S Research, LLC, Miami, Florida
  - The Angel Medical Research Corporation, Miami Lakes, Florida
  - South Florida Research, Miami Springs, Florida
  - EMINAT Research, Miramar, Florida
  - Combined Research Orlando Phase I-IV LLC, Orlando, Florida
  - Ormond Beach Clinical Research, Ormond Beach, Florida
  - CTMD Research, Inc. - Palm Springs - Hunt - PPDS, Palm Springs, Florida
  - IMIC Inc., Palmetto Bay, Florida
  - Infectious Disease Consultants of the Treasure Coast, Sebastian, Florida
  - Westchester General Hospital, South Miami, Florida
  - DBC Research, Tamarac, Florida
  - Alliance Clinical Research-(Tampa), Tampa, Florida
  - Palm Beach Research - ClinEdge - PPDS, West Palm Beach, Florida
  - Agile Clinical Research Trials, LLC, Atlanta, Georgia
  - Centricity Research - Roswell - HyperCore - PPDS, Columbus, Georgia
  - Eagle Clinical Research, Chicago, Illinois
  - Revival Research Corporation - Clinedge - PPDS, Sterling Heights, Michigan
  - Safe Haven Clinical Research, Clinton, Mississippi
  - Mercury Street Medical Group, Butte, Montana
  - Las Vegas Medical Research, Las Vegas, Nevada
  - Research Carolina Elite, Denver, North Carolina
  - WellNow Urgent Care Troy Urgent Care, Dayton, Ohio
  - STAT Research, Vandalia, Ohio
  - Clinovacare Medical Clinical Research Center, West Columbia, South Carolina
  - Veritas Health Care Group, West Columbia, South Carolina
  - Clinical Trials Center of Middle Tennessee, Franklin, Tennessee
  - Central Texas Clinical Research, Austin, Texas
  - Zenos Clinical Research, Dallas, Texas
  - Proactive Clinical Research, LLC Edinburg, Edinburg, Texas
  - Care United Research, LLC, Forney, Texas
  - Mercy Family Clinic, Houston, Texas
  - Xpress Trials, Houston, Texas
  - Diversified Medical Practices, P.A., Houston, Texas
  - Epic Clinical Research, Lewisville, Texas
  - VIP Trials, San Antonio, Texas
  - Suffolk Multispecialty Research, Suffolk, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PBI-0451 (Pomotrelvir) | Placebo
Started | 162 | 80
Completed | 154 | 77
Not Completed | 8 | 3
Not completed — Study drug non-compliance/ | 5 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — concurrent illness | 0 | 1
Not completed — Pregnancy | 1 | 1

BASELINE CHARACTERISTICS:
Population: A blood specimen will be collected for the evaluation of immune biomarkers that could regulate or be involved in the disposition of SARS-CoV-2 or PBI-0451. This sample will be collected @ baseline &SARS-CoV-2 (MT swab) evaluate the potential for PBI-0451resistance development w/additional time points evaluated if virologic rebound or subject remains viremic at other study visits (SARS-CoV-2 RNA by qRT-PCR is ≥ 3.85 log10 copies/mL (meeting min threshold for whole genome sequencing).
Groups:
- Total: Total of all reporting groups
Arm/Group | PBI-0451 (Pomotrelvir) | Placebo | Total
Number analyzed (Participants) | 162 | 80 | 242
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 161 | 79 | 240
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (12.29) | 42.4 (11.75) | 42.6 (12.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 42 | 127
  Male | 77 | 38 | 115
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 162 | 80 | 242

OUTCOME MEASURES:

1. Primary Outcome: Virologic Efficacy of PBI-0451 (Pomotrelvir)
Description: The primary efficacy endpoint was the proportion of participants below LOD for infectious SARS-CoV-2 on Day 3 by IVA from MT nasal swabs for the mITTV analysis set.
Time Frame: Day 3
Population: The mITTV analysis set included a subset of the mITT anaylsis set who had detectable infectious SARS-CoV-2 at baseline/Day 1.
Measure: Count of Participants; unit: Participants
Arm/Group | PBI-0451 (Pomotrelvir) | Placebo
Number analyzed (Participants) | 84 | 39
Participants | 37 | 20

2. Secondary Outcome: Safety and Tolerability of PBI-0451(Pomotrelvir)
Description: Number of treatment-emergent adverse events (AEs), serious adverse events (SAEs), discontinuations due to AEs, and Grade 3 or 4 laboratory abnormalities
Time Frame: Day 1-28
Population: The safety analysis set included all randomized participants who received ≥ 1 dose of study drug.
Measure: Number; unit: events
Arm/Group | PBI-0451 (Pomotrelvir) | Placebo
Number analyzed (Participants) | 161 | 80
events
  Adverse Events | 26 | 4
  Serious Adverse Events | 1 | 0
  Discontinuation of study drug due to AEs | 1 | 0
  Grade 3 Lab Abnormalities | 15 | 4
  Grade 4 Lab Abnormalities | 1 | 3

3. Secondary Outcome: Clinical Efficacy of PBI-0451(Pomotrelvir) Versus Placebo Through Study Day 28
Description: Number of Pomotrelvir treated participants with sustained symptom resolution through Day 28 versus untreated Placebo participants
Time Frame: Day 1 - 28
Population: Participants who met sustained resolution of symptoms through Day 28
Measure: Number; unit: participants
Arm/Group | PBI-0451 (Pomotrelvir) | Placebo
Number analyzed (Participants) | 153 | 77
participants | 132 | 66

4. Secondary Outcome: Effect of PBI-0451(Pomotrelvir) on SARS-CoV-2
Description: Presence of SARS-CoV-2 virus, viral RNA or viral antigen based on IVA, quantitative reverse transcriptase polymerase chain reaction (qRT-PCR), and rapid antigen test (RAT), as specified in the Clinical Virology Analysis Plan (CVAP)
Time Frame: Day 1-28
Population: Numbers reflect subjects with sufficient viral load at baselline for whole genome sequencing.
Measure: Count of Participants; unit: Participants
Arm/Group | PBI-0451 (Pomotrelvir) | Placebo
Number analyzed (Participants) | 53 | 32
Participants | 37 | 20

5. Secondary Outcome: Clinical Efficacy of PBI-0451(Pomotrelvir) Versus Placebo Through Study Day 1-28
Description: The median number of days to sustained resolution of of all 14 COVID-19 symptoms for the PBI-0451 vs Placebo groups through Day 28.
Time Frame: Day 1-28
Population: The median number of days to cessation of 14 targeted CVOID-19 symptoms reported at baseline.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | PBI-0451 (Pomotrelvir) | Placebo
Number analyzed (Participants) | 153 | 77
days | 10 [8 to 11] | 11 [8 to 11]

6. Other Pre Specified Outcome: Incidence of Rebound SARS-CoV-2 Infection
Description: Percentage of participantss with clinical and/or virologic rebound
Time Frame: Day 1-28
Measure: Count of Participants; unit: Participants
Arm/Group | PBI-0451 (Pomotrelvir) | Placebo
Number analyzed (Participants) | 153 | 77
Participants | 14 | 2

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | PBI-0451 (Pomotrelvir) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/162 | 0/80
Serious Adverse Events (participants affected / at risk) | 1/162 | 0/80
Other Adverse Events (participants affected / at risk) | 22/162 | 4/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PBI-0451 (Pomotrelvir) (N=162) | Placebo (N=80)
hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PBI-0451 (Pomotrelvir) (N=162) | Placebo (N=80)
Nausea (Gastrointestinal disorders) | 7 (7) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 2 (2) | 0 (0)
Urinaryl tract infection (Renal and urinary disorders) | 2 (2) | 0 (0)
Dysgeusia (General disorders) | 2 (2) | 0 (0)
other GI (Gastrointestinal disorders) | 2 (2) | 3 (3)
other infection (Infections and infestations) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-10): https://cdn.clinicaltrials.gov/large-docs/07/NCT05543707/Prot_SAP_001.pdf